CLINICAL TRIAL: NCT00622232
Title: A Rollover Study to Evaluate Safety and Therapeutic Effect of Re-infusing Subjects Who Completed Participation in the VRX496-USA-05-002 Trial With Autologous T Cells Transduced With VRX496
Brief Title: A Rollover Study for Subjects Who Completed Participation in the VRX496-USA-05-002 Trial
Acronym: Rollover
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VIRxSYS Corporation (Industry)
Responsible Party: Tessio Rebello, PhD/Vice President of Clinical Affairs, VIRxSYS Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRX496-USA-05-002-Rollover
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV-1; treatment experienced, complementary therapies
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: VRX496-transduced autologous CD4 T cells — The cell dose will consist of approximately 10 billion VRX496-transduced autologous CD4 T cells provided as a single bolus infusion.

SUMMARY:
The objective of this study is to determine the long term safety and tolerability of an additional infusion of 10 billion VRX496 gene-modified CD4 T cells with a focus on evaluating additional therapeutic benefits with respect to viral load and CD4 counts.

DETAILED DESCRIPTION:
The study has concluded it's 9-month active phase. Subjects are currently in a 15-year Long Term Follow-up Phase of the study.

In keeping with the recently released Guidance on Monitoring For Delayed Adverse Events, that states that for the first 5 years all subjects should undergo monitoring of vector sequences every 6 months, subjects will visit the clinic at a maximum of 6 months intervals for a blood test evaluating persistence of vector sequences.

Therefore for the first 5 years, subjects will have 6 months visits for safety assessment. For years 6 to 15, subjects will be contacted by phone or mail. At these contacts, subjects will be asked about their health status.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written informed consent in accordance with institutional and federal guidelines and to comply with the investigational nature of the study and the related requirements.
* Subjects who have successfully completed participation in the VRX496-USA-05-002 trial.
* Subjects who initiated or changed to a new ARV regimen more than 3 months prior to Entry Assessment are eligible.
* Subjects that who (1) if on ARVs and are willing to continue on the current therapy unchanged, or (2) if not on ARV willing to remain off ARVs for the duration of the trial i.e. 9 months. However, if there is clinical need to start or change ARV therapy, then it is permitted to do so.

Exclusion Criteria:

* CD4 counts decreased by ≥25% from baseline in main study.
* Viral load increased by ≥ 1.0 log from baseline in main study or ≥ 200,000.
* Female subjects who are of reproductive potential who have a positive serum B HCG at the Entry Assessment visit or are not willing to use a reliable method of barrier contraception.
* Are breast-feeding.
* Subjects who are actively using injection drugs or other substance abuse (such as extensive alcohol or narcotic use).
* Any medical condition(s) which, in the opinion of the investigator, would interfere with the subject's ability to participate in or adhere to the requirements of this protocol
* Active HIV-related or non HIV-related illness
* Subjects who do not have additional cell product available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of an additional infusion of VRX496 CD4+ T cells in subjects who previously received VRX496 CD4 T cells under protocol VRX496-USA-05-002. | 9 months
To evaluate the change in log10 HIV-1 RNA level | 9 months
To evaluate the change between main study baseline CD4 counts and Month 9 post reinfusion | 9 months

SECONDARY OUTCOMES:
Changes in immune function as determined by ICS and TCR vβ Repertoire profile. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Tessio E Rebello, PhD, Study Director — VIRxSYS Corporation; David Stein, M.D., Principal Investigator — Jacobi Medical Center; Gary Blick, M.D., Principal Investigator — CIRCLE Medical, LLC
Locations (2):
- United States (2):
  - CIRCLE Medical, LLC, Norwalk, Connecticut
  - Jacobi Medical Center, New York, New York